CLINICAL TRIAL: NCT03800030
Title: A Pilot Study Investigating the Effects of Cross Frequency Transcranial Alternating Current Stimulation on Cortical Oscillations Underlying Cognition
Brief Title: Effect of Cross Frequency tACS on Cognitive Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 18-0003; R01MH101547 (NIH)
Record Dates: First submitted 2018-12-18; First posted 2019-01-10 (Actual); Results first posted 2020-05-18 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2019-09

CONDITIONS: Cognitive Control; Executive Function
Keywords: tACS; Cognitive Control; Executive Function

STUDY DESIGN:
Intervention Model Description: Healthy participants will receive three waveforms of transcranial alternating current stimulation (tACS). Delta-beta, Theta-gamma, and Sham.
Who Masked: Participant, Investigator
Masking Description: Double-blinded. Neither the investigator nor the participants knows which form of stimulation is received.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Theta-gamma, Delta-beta, Sham (Experimental): Every participant will receive Theta-gamma tACS, Delta-beta tACS, and Sham tACS on separate sessions during performance of a computerized task.
  Sequence: Theta-gamma tACS, then Delta-beta tACS, then Sham tACS
  Interventions: Device: Theta-gamma tACS; Device: Delta-beta tACS; Device: Sham tACS
- Theta-gamma, Sham, Delta-beta (Experimental): Every participant will receive Theta-gamma tACS, Delta-beta tACS, and Sham tACS on separate sessions during performance of a computerized task.
  Sequence: Theta-gamma tACS, then Sham tACS, then Delta-beta tACS
  Interventions: Device: Theta-gamma tACS; Device: Delta-beta tACS; Device: Sham tACS
- Delta-beta, Theta-gamma, Sham tACS (Experimental): Every participant will receive Theta-gamma tACS, Delta-beta tACS, and Sham tACS on separate sessions during performance of a computerized task.
  Sequence: Delta-beta tACS, then Theta-gamma tACS, then Sham tACS
  Interventions: Device: Theta-gamma tACS; Device: Delta-beta tACS; Device: Sham tACS
- Delta-beta, Sham, Theta-gamma tACS (Experimental): Every participant will receive Theta-gamma tACS, Delta-beta tACS, and Sham tACS on separate sessions during performance of a computerized task.
  Sequence: Delta-beta tACS, then Sham tACS, then Theta-gamma tACS
  Interventions: Device: Theta-gamma tACS; Device: Delta-beta tACS; Device: Sham tACS
- Sham, Delta-beta, Theta-gamma tACS (Experimental): Every participant will receive Theta-gamma tACS, Delta-beta tACS, and Sham tACS on separate sessions during performance of a computerized task.
  Sequence: Sham tACS, then Delta-beta tACS, then Theta-gamma tACS
  Interventions: Device: Theta-gamma tACS; Device: Delta-beta tACS; Device: Sham tACS
- Sham, Theta-gamma, Delta-beta tACS (Experimental): Every participant will receive Theta-gamma tACS, Delta-beta tACS, and Sham tACS on separate sessions during performance of a computerized task.
  Sequence: Sham tACS, then Theta-gamma tACS, then Delta-beta tACS
  Interventions: Device: Theta-gamma tACS; Device: Delta-beta tACS; Device: Sham tACS

INTERVENTIONS:
Device: Theta-gamma tACS — NeuroConn technologies, direct current-stimulator plus
Device: Delta-beta tACS — NeuroConn technologies, direct current-stimulator plus
Device: Sham tACS — NeuroConn technologies, direct current-stimulator plus

SUMMARY:
Investigation of frequency specific transcranial alternating current stimulation on cognitive control signals in frontal cortex

DETAILED DESCRIPTION:
Previous evidence suggests that there are specific frequency bands associated with different aspects of cognitive control. In specific delta (2-4Hz) and beta (15-30Hz) are associated with increased levels of abstraction for learned rules; and theta (5-8Hz) and gamma (30-50Hz) has been associated with increased set-size or number of learned rules. Here we aim to find causal evidence in support of these previous correlational findings by applying cross-frequency transcranial alternating current stimulation (tACS) in the specific frequency bands previously shown to be task-relevant. In a crossover design, we stimulate subjects with either delta-beta or theta-gamma tACS during performance of a hierarchical cognitive control task that manipulates the level of abstraction and set-size of rules that must be learned in order to make the correct button press.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 35 years
* Able to provide informed consent
* Willing to comply with all study procedures and be available for the duration of the study Speak and understand English

Exclusion Criteria:

* Attention Deficit Hyperactivity Disorder (currently under treatment)
* Neurological disorders and conditions, including, but not limited to:
* History of epilepsy
* Seizures (except childhood febrile seizures and electroconvulsive therapy induced seizures) Dementia
* History of stroke
* Parkinson's disease
* Multiple sclerosis
* Cerebral aneurysm
* Brain tumors
* Medical or neurological illness or treatment for a medical disorder that could interfere with study participation (e.g., unstable cardiac disease, malignancy)
* Prior brain surgery
* Any brain devices/implants, including cochlear implants and aneurysm clips
* History or current traumatic brain injury
* (For females) Pregnancy or breast feeding
* Personal or family history of mental/psychiatric disorder (e.g., anxiety, major depressive disorder, schizophrenia, etc.)
* Positive urine test for the following: Marijuana (THC), Cocaine (COC), Phencyclidine (PCP), Amphetamine (AMP), Ecstasy (MDMA), Methamphetamine (Mamp), Opiates (OPI), Oxycodone (OXY), Methadone (MTD), Barbiturates (BAR), Benzodiazepines (BZO), Buprenorphine (BUP), Tricyclic Antidepressants (TCA), Propoxyphene (PPX)
* Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-10-07 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Riddle J, McFerren A, Frohlich F. Causal role of cross-frequency coupling in distinct components of cognitive control. Prog Neurobiol. 2021 Jul;202:102033. doi: 10.1016/j.pneurobio.2021.102033. Epub 2021 Mar 16. PMID 33741402

RESULTS

PARTICIPANT FLOW:
Groups:
- Theta-gamma, Delta-beta, Sham: Every participant will receive Theta-gamma tACS, Delta-beta tACS, and Sham tACS on separate sessions during performance of a computerized task.
  Sequence: Theta-gamma tACS, then Delta-beta tACS, then Sham tACS
  Theta-gamma tACS: NeuroConn technologies, direct current-stimulator plus
  Delta-beta tACS: NeuroConn technologies, direct current-stimulator plus
  Sham tACS: NeuroConn technologies, direct current-stimulator plus
- Theta-gamma, Sham, Delta-beta: Every participant will receive Theta-gamma tACS, Delta-beta tACS, and Sham tACS on separate sessions during performance of a computerized task.
  Sequence: Theta-gamma tACS, then Sham tACS, then Delta-beta tACS
  Theta-gamma tACS: NeuroConn technologies, direct current-stimulator plus
  Delta-beta tACS: NeuroConn technologies, direct current-stimulator plus
  Sham tACS: NeuroConn technologies, direct current-stimulator plus
- Delta-beta, Theta-gamma, Sham tACS: Every participant will receive Theta-gamma tACS, Delta-beta tACS, and Sham tACS on separate sessions during performance of a computerized task.
  Sequence: Delta-beta tACS, then Theta-gamma tACS, then Sham tACS
  Theta-gamma tACS: NeuroConn technologies, direct current-stimulator plus
  Delta-beta tACS: NeuroConn technologies, direct current-stimulator plus
  Sham tACS: NeuroConn technologies, direct current-stimulator plus
- Delta-beta, Sham, Theta-gamma tACS: Every participant will receive Theta-gamma tACS, Delta-beta tACS, and Sham tACS on separate sessions during performance of a computerized task.
  Sequence: Delta-beta tACS, then Sham tACS, then Theta-gamma tACS
  Theta-gamma tACS: NeuroConn technologies, direct current-stimulator plus
  Delta-beta tACS: NeuroConn technologies, direct current-stimulator plus
  Sham tACS: NeuroConn technologies, direct current-stimulator plus
- Sham, Delta-beta, Theta-gamma tACS: Every participant will receive Theta-gamma tACS, Delta-beta tACS, and Sham tACS on separate sessions during performance of a computerized task.
  Sequence: Sham tACS, then Delta-beta tACS, then Theta-gamma tACS
  Theta-gamma tACS: NeuroConn technologies, direct current-stimulator plus
  Delta-beta tACS: NeuroConn technologies, direct current-stimulator plus
  Sham tACS: NeuroConn technologies, direct current-stimulator plus
- Sham, Theta-gamma, Delta-beta tACS: Every participant will receive Theta-gamma tACS, Delta-beta tACS, and Sham tACS on separate sessions during performance of a computerized task.
  Sequence: Sham tACS, then Theta-gamma tACS, then Delta-beta tACS
  Theta-gamma tACS: NeuroConn technologies, direct current-stimulator plus
  Delta-beta tACS: NeuroConn technologies, direct current-stimulator plus
  Sham tACS: NeuroConn technologies, direct current-stimulator plus
Period: Baseline
Arm/Group | Theta-gamma, Delta-beta, Sham | Theta-gamma, Sham, Delta-beta | Delta-beta, Theta-gamma, Sham tACS | Delta-beta, Sham, Theta-gamma tACS | Sham, Delta-beta, Theta-gamma tACS | Sham, Theta-gamma, Delta-beta tACS
Started | 4 | 4 | 4 | 6 | 4 | 4
Completed | 4 | 4 | 4 | 6 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Pre-Randomization Period (1 Week)
Arm/Group | Theta-gamma, Delta-beta, Sham | Theta-gamma, Sham, Delta-beta | Delta-beta, Theta-gamma, Sham tACS | Delta-beta, Sham, Theta-gamma tACS | Sham, Delta-beta, Theta-gamma tACS | Sham, Theta-gamma, Delta-beta tACS
Started | 4 | 4 | 4 | 6 | 4 | 4
Completed | 4 | 4 | 4 | 6 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: First Intervention
Arm/Group | Theta-gamma, Delta-beta, Sham | Theta-gamma, Sham, Delta-beta | Delta-beta, Theta-gamma, Sham tACS | Delta-beta, Sham, Theta-gamma tACS | Sham, Delta-beta, Theta-gamma tACS | Sham, Theta-gamma, Delta-beta tACS
Started | 4 | 4 | 4 | 6 | 4 | 4
Completed | 4 | 4 | 4 | 6 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: First Washout (1 Week)
Arm/Group | Theta-gamma, Delta-beta, Sham | Theta-gamma, Sham, Delta-beta | Delta-beta, Theta-gamma, Sham tACS | Delta-beta, Sham, Theta-gamma tACS | Sham, Delta-beta, Theta-gamma tACS | Sham, Theta-gamma, Delta-beta tACS
Started | 4 | 4 | 4 | 6 | 4 | 4
Completed | 4 | 4 | 4 | 6 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention
Arm/Group | Theta-gamma, Delta-beta, Sham | Theta-gamma, Sham, Delta-beta | Delta-beta, Theta-gamma, Sham tACS | Delta-beta, Sham, Theta-gamma tACS | Sham, Delta-beta, Theta-gamma tACS | Sham, Theta-gamma, Delta-beta tACS
Started | 4 | 4 | 4 | 6 | 4 | 4
Completed | 4 | 4 | 4 | 5 | 4 | 4
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Period: Second Washout (1 Week)
Arm/Group | Theta-gamma, Delta-beta, Sham | Theta-gamma, Sham, Delta-beta | Delta-beta, Theta-gamma, Sham tACS | Delta-beta, Sham, Theta-gamma tACS | Sham, Delta-beta, Theta-gamma tACS | Sham, Theta-gamma, Delta-beta tACS
Started | 4 | 4 | 4 | 5 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 1 | 0 | 0
Period: Third Intervention
Arm/Group | Theta-gamma, Delta-beta, Sham | Theta-gamma, Sham, Delta-beta | Delta-beta, Theta-gamma, Sham tACS | Delta-beta, Sham, Theta-gamma tACS | Sham, Delta-beta, Theta-gamma tACS | Sham, Theta-gamma, Delta-beta tACS
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Every participant will receive Theta-gamma tACS, Delta-beta tACS, and Sham tACS on separate sessions during performance of a computerized task.
Arm/Group | All Participants
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.654 (1.4951)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 17
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 15
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26
Baseline Reaction Time Difference for Abstraction [Mean (Standard Deviation); unit: seconds] — There are four task conditions in a two-by-two design for high and low set-size and high and low abstraction. The reaction time for both high abstraction conditions are averaged and the average reaction time for both low abstraction conditions is subtracted. Thus, a single reaction metric is derived that is the relative change in reaction time as a function of the abstraction of the task. Population: One participant excluded from behavioral analysis because they did not follow task instructions. Two participants did not complete the full study and thus were excluded from analysis.
  seconds
    number analyzed (Participants) | 23
    (all) | 0.1637 (0.1012)
Baseline Reaction Time Difference for Set-Size [Mean (Standard Deviation); unit: seconds] — There are four task conditions in a two-by-two design for high and low set-size and high and low abstraction. The reaction time for both high set-size conditions are averaged and the average reaction time for both low set-size conditions is subtracted. Thus, a single reaction metric is derived that is the relative change in reaction time as a function of the set-size of the task. Population: One participant excluded from behavioral analysis because they did not follow task instructions. Two participants did not complete the full study and thus were excluded from analysis.
  seconds
    number analyzed (Participants) | 23
    (all) | 0.2272 (0.0844)
Baseline Percent Correct Difference for Abstraction [Mean (Standard Deviation); unit: percent correct] — There are four task conditions in a two-by-two design for high and low set-size and high and low abstraction. The percent correct for both high abstraction conditions are averaged and the average percent correct for both low abstraction conditions is subtracted. Thus, a single metric is derived that is the relative change in percent correct as a function of the abstraction of the task. Population: One participant excluded from behavioral analysis because they did not follow task instructions. Two participants did not complete the full study and thus were excluded from analysis.
  percent correct
    number analyzed (Participants) | 23
    (all) | 0.0679 (4.9692)
Baseline Percent Correct Difference for Set-Size [Mean (Standard Deviation); unit: percent correct] — There are four task conditions in a two-by-two design for high and low set-size and high and low abstraction. The percent correct for both high st-size conditions are averaged and the average percent correct for both low set-size conditions is subtracted. Thus, a single metric is derived that is the relative change in percent correct as a function of the set-size of the task. Population: One participant excluded from behavioral analysis because they did not follow task instructions. Two participants did not complete the full study and thus were excluded from analysis.
  percent correct
    number analyzed (Participants) | 23
    (all) | -1.0190 (4.4569)
Baseline Delta Phase to Beta Amplitude Coupling [Mean (Standard Deviation); unit: Z-score] — During resting-state EEG, the Hilbert transform is applied at delta (2-3 Hz) and beta (18-22 Hz) frequency band. The phase of delta and the amplitude of beta frequency oscillations are combined into a single hybrid signal. Then, this signal is averaged and the magnitude of the resulting vector is taken as the coupling strength. To account for spurious findings, a null distribution is calculated by randomly shifting the time series of amplitude values. The final coupling measure is z-transformed by subtracting the mean and dividing by the standard deviation of the null distribution. Population: One participant excluded from behavioral analysis because they did not follow task instructions. Two participants did not complete the full study and thus were excluded from analysis.
  Z-score
    number analyzed (Participants) | 23
    (all) | 0.0406 (0.3232)
Theta Phase to Gamma Amplitude Coupling Strength [Mean (Standard Deviation); unit: Z-score] — During resting-state EEG, the Hilbert transform is applied at theta (4-8 Hz) and gamma (30-50 Hz) frequency band. The phase of theta and the amplitude of gamma frequency oscillations are combined into a single hybrid signal. Then, this signal is averaged and the magnitude of the resulting vector is taken as the coupling strength. To account for spurious findings, a null distribution is calculated by randomly shifting the time series of amplitude values. The final coupling measure is z-transformed by subtracting the mean and dividing by the standard deviation of the null distribution. Population: One participant excluded from behavioral analysis because they did not follow task instructions. Two participants did not complete the full study and thus were excluded from analysis.
  Z-score
    number analyzed (Participants) | 23
    (all) | 0.0739 (0.4214)

OUTCOME MEASURES:

1. Primary Outcome: Reaction Time for Trials With High Abstraction Relative to Low Abstraction
Description: For low abstraction conditions, subjects must memorize a color to button mapping. For high abstraction conditions, subject must make a perceptual judgement on the similarity of two objects based on either texture or shape as cued by a color. The reaction time difference between high and low abstraction conditions was hypothesized to decrease when delta-beta tACS was delivered. As a control for the placebo effect of stimulation, the difference between delta-beta tACS and sham tACS, or placebo, was used for statistical analysis.
Time Frame: through study completion, an average of 3 weeks
Population: One participant excluded from behavioral analysis because they did not follow task instructions.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Theta-gamma tACS: Every participant will receive Theta-gamma tACS during performance of a computerized task using NeuroConn technologies, direct current-stimulator plus
- Delta-beta tACS: Every participant will receive Delta-beta tACS during performance of a computerized task using NeuroConn technologies, direct current-stimulator plus
- Sham tACS: Every participant will receive Sham tACS during performance of a computerized task using NeuroConn technologies, direct current-stimulator plus
Arm/Group | Theta-gamma tACS | Delta-beta tACS | Sham tACS
Number analyzed (Participants) | 23 | 23 | 23
seconds | 0.1247 (0.0800) | 0.1444 (0.0832) | 0.1022 (0.0947)
Statistical Analysis 1: Comparison: Delta-beta tACS vs Sham tACS; Test type: Superiority; p = 0.031, t-test, 2 sided; degrees of freedom = 22 t-statistic = 2.305

2. Primary Outcome: Reaction Time for Trials With High Set-size Relative to Low Set-size
Description: The reaction time difference between high and low set-size conditions was hypothesized to decrease when theta-gamma tACS is delivered. As a control for the placebo effect of stimulation, the difference between theta-gamma tACS and sham tACS, or placebo, was used for statistical analysis.
Time Frame: through study completion, an average of 3 weeks
Population: One participant excluded from behavioral analysis because they did not follow task instructions.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Theta-gamma tACS | Delta-beta tACS | Sham tACS
Number analyzed (Participants) | 23 | 23 | 23
seconds | 0.1905 (0.0676) | 0.1853 (0.1057) | 0.1888 (0.0760)
Statistical Analysis 1: Comparison: Theta-gamma tACS vs Sham tACS; Test type: Superiority; p = 0.935, t-test, 2 sided; degrees of freedom = 22 t-statistic = 0.083

3. Primary Outcome: Delta Phase to Beta Amplitude Coupling Strength
Description: Delta-beta tACS was hypothesized to increase cross frequency coupling strength (higher value) between the targeted frequency bands. Phase amplitude coupling between delta phase and beta amplitude was calculated for the two minute electrical brain recordings after stimulation. A null distribution was calculated by shuffling the beta amplitude time series relative to the delta phase time series and then calculating coupling strength. The outcome measure is the z-transformed value of the genuine phase amplitude coupling relative to the null distribution.
Time Frame: through study completion, an average of 3 weeks
Population: One participant excluded from coupling analysis because they did not follow task instructions.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Theta-gamma tACS | Delta-beta tACS | Sham tACS
Number analyzed (Participants) | 23 | 23 | 23
Z-score | -0.0873 (0.3035) | 0.1123 (0.2939) | -0.1250 (0.2651)
Statistical Analysis 1: Comparison: Theta-gamma tACS vs Delta-beta tACS vs Sham tACS; Test type: Superiority; p = 0.040, t-test, 1 sided; degrees of freedom = 22 t-statistic = 1.833

4. Primary Outcome: Theta Phase to Gamma Amplitude Coupling Strength
Description: Theta-gamma tACS was hypothesized to increase cross frequency coupling strength (higher value) between the targeted frequency bands. Phase amplitude coupling between theta phase and gamma amplitude was calculated for the two minute electrical brain recordings after stimulation. A null distribution was calculated by shuffling the gamma amplitude time series relative to the theta phase time series and then calculating coupling strength. The outcome measure is the z-transformed value of the genuine phase amplitude coupling relative to the null distribution.
Time Frame: through study completion, an average of 3 weeks
Population: One participant was excluded from coupling analysis because they did not follow task instructions.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Theta-gamma tACS | Delta-beta tACS | Sham tACS
Number analyzed (Participants) | 23 | 23 | 23
Z-score | 0.1615 (0.3563) | 0.0706 (0.3496) | 0.0577 (0.4043)
Statistical Analysis 1: Comparison: Theta-gamma tACS vs Sham tACS; Test type: Superiority; p = 0.020, t-test, 1 sided; degrees of freedom = 22 t-statistic = 2.174

5. Primary Outcome: Percent Correct for Trials With High Abstraction Relative to Low Abstraction
Description: For low abstraction conditions, subjects must memorize a color to button mapping. For high abstraction conditions, subject must make a perceptual judgement on the similarity of two objects based on either texture or shape as cued by a color. The accuracy difference between high and low abstraction conditions was hypothesized to decrease when delta-beta tACS was delivered. As a control for the placebo effect of stimulation, the difference between delta-beta tACS and sham tACS, or placebo, was used for statistical analysis.
Time Frame: through study completion, an average of 3 weeks
Population: One participant excluded from behavioral analysis because they did not follow task instructions.
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Theta-gamma tACS | Delta-beta tACS | Sham tACS
Number analyzed (Participants) | 23 | 23 | 23
percent correct | 0.5661 (3.1678) | -0.2944 (7.4718) | 0.7246 (6.6416)
Statistical Analysis 1: Comparison: Delta-beta tACS vs Sham tACS; Test type: Superiority; p = 0.540, t-test, 2 sided; degrees of freedom = 22 t-statistic = -0.623

6. Primary Outcome: Percent Correct for Trials With High Set-size Relative to Low Set-size
Description: The accuracy difference between high and low set-size conditions was hypothesized to decrease when theta-gamma tACS is delivered. As a control for the placebo effect of stimulation, the difference between theta-gamma tACS and sham tACS, or placebo, was used for statistical analysis.
Time Frame: through study completion, an average of 3 weeks
Population: One participant excluded from behavioral analysis because they did not follow task instructions.
Measure: Mean (Standard Deviation); unit: percent correct
Arm/Group | Theta-gamma tACS | Delta-beta tACS | Sham tACS
Number analyzed (Participants) | 23 | 23 | 23
percent correct | -2.2871 (2.9242) | -4.3252 (6.8997) | -4.1667 (4.3264)
Statistical Analysis 1: Comparison: Theta-gamma tACS vs Sham tACS; Test type: Superiority; p = 0.007, t-test, 2 sided; degrees of freedom = 22 t-statistic = 2.989

ADVERSE EVENTS:
Time Frame: Adverse events were assessed over an approximate 3-week period using a stimulation side effects questionnaire provided to participants after every presentation of each intervention. Data were not collected beyond the third intervention.
Arm/Group | Theta-gamma tACS | Delta-beta tACS | Sham tACS
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 11/24 | 15/26 | 10/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Theta-gamma tACS (N=24) | Delta-beta tACS (N=26) | Sham tACS (N=26)
Tingling (Investigations) | 9 (9) | 10 (10) | 7 (7) — Mild
Flickering lights (Investigations) | 2 (2) | 4 (4) | 2 (2) — Mild
Itching (Investigations) | 2 (2) | 5 (5) | 4 (4) — Mild
Burning sensation (Investigations) | 3 (3) | 3 (3) | 5 (5) — Mild
Scalp pain (Investigations) | 3 (3) | 3 (3) | 2 (2) — Mild
Neck pain (Investigations) | 1 (1) | 1 (1) | 0 (0) — Mild
Dizziness (Investigations) | 0 (0) | 3 (3) | 0 (0) — Mild
Local redness (Investigations) | 1 (1) | 1 (1) | 0 (0) — Mild
Sleepiness (Investigations) | 1 (1) | 0 (0) | 0 (0) — Mild
Headache (Investigations) | 3 (3) | 1 (1) | 3 (3) — Mild
Ringing noise (Investigations) | 1 (1) | 0 (0) | 0 (0) — Mild
Blurred vision (Investigations) | 0 (0) | 0 (0) | 1 (1) — Mild

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT03800030/Prot_SAP_000.pdf